CLINICAL TRIAL: NCT05147623
Title: Postoperative Mortality in Colombia: Perspectives of the Fourth Indicator in The Lancet Commission on Global Surgery (Colombian Surgical Outcomes Study)
Brief Title: Colombian Surgical Outcomes Study - COLSOS
Acronym: COLSOS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundación Cardioinfantil Instituto de Cardiología (Other)
Collaborators: Universidad del Rosario (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-PRO-CAR-1538
Record Dates: First submitted 2021-11-24; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Surgery; Postoperative Complications; Hospital Mortality
Keywords: Hospital mortality; Postoperative complications; Surgery; Public Health
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Principal cohort: All patients recruited in one week who underwent to any surgical procedure that meet inclusion criteria of the study.
  Interventions: Procedure: Any surgery/procedure

INTERVENTIONS:
Procedure: Any surgery/procedure — Any surgery/procedure in all adult patients that were performed in an operating room

SUMMARY:
An observational, analytical, multicentre prospective cohort study will be conducted throughout Colombia. A sample size of 1353 patients is needed to achieve significance in our primary objective; however, convenience sampling is considered, as we aim to include all the institutions and patients possible. The data collection will be carried out prospectively for one week, and all patients will have a follow-up of a maximum of 30 days in-hospital. The primary outcome will be to determine the in-hospital mortality. We aim to contribute with accurate information on in-hospital postoperative mortality in Colombia. Thus, by following precisely the instructions created by The Lancet Commission on Global Surgery. The data obtained will help formulate public policies in the surgical field adjusted to the Colombian population, improving the quality of the surgical divisions in the different Colombian institutions, positively affecting the attention and development of the Colombian healthcare system.

DETAILED DESCRIPTION:
The general objective of this research is to describe the in-hospital postoperative mortality of patients who have had surgical procedures in Colombian institutions.

We also aim to characterize the sociodemographic and clinical variables of the patients that underwent a surgical procedure in Colombia, determine the secondary postoperative clinical outcomes associated with surgical procedures in Colombia and illustrate the installed surgical capacity and infrastructure of the participating health centres.

The study will be carried out throughout Colombia. The largest number possible of institutions in which surgeries are performed will be included. We expect to have at least 2 or 3 institutions per region. We currently have 65 confirmed participating institutions and have conducted a preliminary interaction with 257 institutions throughout the territory. The list of participating centres and researchers will be continuously updated, and the final version of the list will be attached to the final report.

A sample size estimate of 1353 patients was made to establish the lower limit needed to achieve significance in our primary objective. The estimate was made with the postoperative mortality rate in Colombia obtained in the study by Hanna et al. of 0.74% (13), an alpha value of 0.05, an accuracy of 0.5%, and a design effect of 1.2. Also, due to the nature of the study, it is not possible to randomize. Nevertheless, convenience sampling is considered, as we aim to include all the patients possible.

A descriptive analysis of the data will be performed. The continuous variables will be assessed whit normality tests (Shapiro Wilk or Kolmogorov Smirnov). If the variables have a normal distribution, they will be expressed as mean (measure of central tendency) and as standard deviation (measure of dispersion). Contrariwise, if the variables have a non-normal distribution, they will be expressed as median (measure of central tendency) and as interquartile range (measure of dispersion).

The continuous data with normal distribution will be studied with parametric tests according to the number of comparators: we will use the student t-test or ANOVA if a comparison of more than two groups is required. For continuous data with non-normal distribution, non-parametric tests will be used: if two groups are compared, we will use the Mann Whitney test, and between three groups, the Kruskal Wallis test. The P-value shall be considered statistically significant < 0,05. Categorical variables shall be presented with absolute frequencies and proportions. Categorical data will be compared between two groups using the Chi-square test or fisher's test at convenience to obtain data after collection.

Logistic regression will be carried out multilevel by individual, city or municipality, department, and country. It will evaluate the association between risk factors and primary outcomes and adjust for differences in confounding factors. A multivariate logistic model will be created for specific mortality comparisons that include all potential risk factors associated with in-hospital mortality. The possible risk factors variables with a variance inflation factor more significant than two were excluded to avoid collinearity.

Four strategies are proposed to attract interested researchers and institutions to participate in this study. Because of the support of the Colombian Surgical Association through the official mail of the organization, a generalized invitation will be sent to all clinics and hospitals with surgical processes, throughout the country, with general information of the research study to attract interest from these institutions. Additionally, the journal and website of the Colombian Surgical Association in both the journal and on the website of the society of general surgery the registration will be published so students, interns, doctors, residents, and specialists interested in participating. Finally, voice-to-voice communication and mass dissemination through ColombianSurg Collaborative social networks (Instagram, Twitter, Facebook, and Official Website) cannot be ruled out.

Coordination with institutions and departments: A hierarchical management organization was set up to generate specific and personalized attention to each region and institution (Figure 3). In addition, researchers will be able to communicate with the ColombianSurg Collaborative team and vice versa through different platforms that will be put at their services, such as instant messaging groups, email, and official Websites.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Ones who underwent to a surgical intervention in the collection period, by the participating institutions.
* Both public and private institutions will be included.
* Patients with and without COVID-19 infection will be included.

Exclusion Criteria:

* Patients who do not have the necessary clinical records to complete the information during data collection.
* Patients who do not approve inclusion in the study through informed consent.
* The following shall be excluded:
* Procedures that were performed outside of operating rooms.
* Radiological procedures.
* Endoscopic procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients of legal age who underwent to surgical procedures by the participating institutions in the data collection period will be included.
Sampling Method: Non-Probability Sample
Enrollment: 1353 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-05-16 (Estimated); Study Completion 2023-05-22 (Estimated)

PRIMARY OUTCOMES:
In-hospital postoperative mortality | 30 days
  In-hospital postoperative mortality of patients who have had surgical procedures in Colombian institutions.

SECONDARY OUTCOMES:
Postoperative complications | 30 days
  Early complications related to surgical procedures that occurred in the selected patients

CONTACTS AND LOCATIONS:
Overall Officials: Paulo A. Cabrera, MD, MSc, Principal Investigator — Fundación Cardioinfantil Instituto de Cardiología; Carlos J. Perez, MD, MSc, Principal Investigator — Fundación Cardioinfantil Instituto de Cardiología
Locations (2):
- Colombia (2):
  - Fundación Cardioinfantil Instituto de Cardiología, Bogotá, Cundinamarca
  - Clínica Avidanti, Ibagué, Tolima Department

IPD SHARING:
Plan to Share IPD: No
The data will be collected and stored online through the server Research Electronic Data Capture(Redcap) web application.
  Redcap allows collaborators to enter data and store it in a security system. The designated collaborator of each hospital will receive the login data in the Redcap system (login), so that the data is sent securely to the server. Only anonymous data will be uploaded to the database. No data will be collected to identify patients. The points of adherence to the STROBE statement have been respected for the study design.

REFERENCES:
- [Derived] Perez-Rivera CJ, Lozano-Suarez N, Velandia-Sanchez A, Polania-Sandoval CA, Garcia-Mendez JP, Idarraga-Ayala SV, Corso-Ramirez JM, Conde-Monroy D, Cruz-Reyes DL, Duran-Torres CF, Barrera-Carvajal JG, Rojas-Serrano LF, Garcia-Zambrano LA, Agudelo-Mendoza SV, Briceno-Ayala L, Cabrera-Rivera PA; ColombianSurg Collaborative. Perioperative mortality in Colombia: perspectives of the fourth indicator in The Lancet Commission on Global Surgery - Colombian Surgical Outcomes Study (ColSOS) - a protocol for a multicentre prospective cohort study. BMJ Open. 2022 Nov 30;12(11):e063182. doi: 10.1136/bmjopen-2022-063182. PMID 36450427